

# Clinical Study Protocol Evaluation of Effectiveness of a Novel Remineralizing Agent: A Randomized Controlled Clinical Trial

| Study Title | Evaluation of Effectiveness of a Novel Remineralizing Agent: A Randomized Controlled Clinical Trial |
|---|---|
| Registration | https://clinicaltrials.gov |
| Study-ID | IVAG-Study-ID: LL4406332<br>Institution-Study-ID: N/A |
| Product | Experimental Fluoride Application |
| Project Number | 62 13 06 |
| Document-ID | LL4470462 |
| Document Version | 1.0 |
| Document Date | 21.03.2022 |

| Document Control | | |
|---|---|---|
| Name | Date | Signature |
| Study Coordinator | 01 -5 0: 40 | |
| Mutlu Özcan | 06.05.2022 | |
| Prof. Dr. Dr. h.c., Ph.D, | | |
| University of Zurich Division of Dental Biomaterials | | |
| Center of Dental Medicine | | |
| Clinic of Reconstructive Dentistry | | |
| Plattenstrasse 11, CH-8032, Zurich, Switzerland | | |
| Mobile: | | |
| E-mail: | | |

| Revision History | | | |
|---|---|---|---|
| Version | Date | Author | Remark on Amendments to the CIP |
| 1.0 | 21.03.2022 | Burcu Gözetici Çil<br>Mutlu Özcan | Initial creation |

#### Evaluation of Effectiveness of a Novel Remineralizing Agent: A Randomized Controlled Clinical Trial



The Coordinating Investigator has approved the CIP version [1.0 (dated 21.03.22), and confirm hereby to conduct the investigation according to the CIP, the current version of the World Medical Association Declaration of Helsinki, ISO14155 norm, ICH-GCP as far as applicable, and the local legally binding requirements. This includes in particular that the clinical investigation shall not begin until the required approval(s) have been obtained and that any additional requirements imposed by the EC or NCA shall be followed, if appropriate.



## **SPONSOR SIGNATURE PAGE**

We, the undersigned, have read this protocol and agree that it contains all necessary information required to conduct the study.

### **Ivoclar Vivadent AG**

Bendererstrasse 2, 9494 Schaan

Liechtenstein



Patrik Oehri

Senior Director CQM & Regulatory Affairs, PRRC



Dr. Thomas Völkel Head of Department Scientific Services / Deputy PRRC Study Management



#### INVESTIGATOR STATEMENT

I have read protocol and agree that it contains all necessary details for carrying out the study described and in conformance with Good Clinical Practices (GCPs), the current version of the World Medical Association Declaration of Helsinki, ISO14155 norm and applicable regulatory requirements. I agree to maintain the confidentiality of all information received or developed in connection with the protocol.

| | - 11 | |
|---------|------|-------|
| RILECTI | GOZO | |
| Burcu | GUZE | |
| | | <br>3 |

Printed Name of Investigator

Signature of Investigator

12,05,2022

Date



# 1. Synopsis

| Sponsor/<br>Manufacturer | Ivoclar Vivadent AG Bendererstrasse 2 9494 Schaan Fürstentum Liechtenstein |
|---|---|
| Study Title | Evaluation of Effectiveness of a Novel Remineralizing Agent: A Randomized Controlled Clinical Trial |
| Short Title | n.a. |
| Version/ Date | 1.0/ 21.03.22 |
| Registration: | https://clinicaltrials.gov |
| Clinical investigation category and Rationale | Medical Device Clinical Trial |
| Background and Rationale: | Active non-cavitated caries lesions on buccal surfaces teeth scored with ICDAS code 1 or 2 are characterized by white chalky appearance as a result of loss of minerals from the tooth structure. The progression of these lesions can be reversed or arrested by application of some therapeutic agents, enhancing remineralization. Fluoride varnishes are considered to be the first choice of treatment for this purpose. Fluoride varnishes with high concentration of fluoride provides calcium fluoride formation which acts as a reservoir for both calcium and fluoride. The release of these ions during acidic challenges inhibits further dissolution of hydroxyapatite crystals of the dental hard tissues. In the present pilot clinical study, the test material containing calcium fluoride nanosol in addition to high level of ammonium fluoride content will be evaluated. Ammonium fluoride solution and calcium fluoride solutions are designed to be applied separately to form a protective layer. Application of calcium fluoride in combination with high concentration of fluoride is anticipated to have beneficial effects on the repair of incipient caries lesions with ICDAS code 1 and 2. |
| Objective(s): | Comparison between investigational medical device (Exp. Fluoride Appl. Ivoclar-Vivadent AG, Schaan, LI) and control product (Fluor Protector S, Ivoclar-Vivadent AG, Schaan, LIE) |
| Outcome(s): | Primary outcome: |



| | <ul> <li>Evaluation of the change in lesion size and mineral content based on Qraycam measurements at baseline, after 1, 6 and 12 months.</li> <li>Secondary outcome: <ul> <li>Clinical evaluation of the lesion progression according to ICDAS and Nyvad criteria at baseline, 1, 6 and 12 months.</li> </ul> </li> <li>Digital pictures for secondary evaluation by the observers to calculate inter-examiner reliability.</li> </ul> |
|---|---|
| Clinical investigation design: | Randomized controlled blinded evaluation in split-mouth design |
| Inclusion / Exclusion criteria: | At least two early caries lesions (arrested or progressive) on buccal sides of two teeth in two different quadrants. Inclusion criteria: Subjects are required to have at least two active non-cavitated white spot lesions (WSLs) on buccal surfaces of anterior teeth or premolars (ICDAS code 1 and 2; Nyvad score 1) Age between 13 and 50 years No untreated caries lesions or periodontal disease No systematic disease or medication (such as antidepressants, antibiotics etc.) that affects salivary flow rate Subjects claimed regular brushing at least twice a day Subjects had to agree to keep the scheduled recall appointments for 1 year. Exclusion criteria: Inactive non-cavitated lesions (Nyvad Score 4) Lesions with microcavity, cavitation, chipping or discoloration Lesions at buccal side of the molars Lesions adjacent to restoration Developmental white spot lesions such as enamel hypoplasia |



| | Pregnant and breastfeeding women |
|---|---|
| | • I regnant and breastreeding women |
| Intervention:<br>Measurements and<br>procedures | The investigational medical device Experimental Fluoride Application, consists of an aqueous fluoride solution and an ethanol-based solution of calcium fluoride nanosol, which is supplied in two separate bottles which will be applied directly on enamel. |
| Control Intervention (if applicable): | Fluor Protector S (Ivoclar Vivadent AG, Schaan, Liechtenstein) is a protective varnish containing ammonium fluoride. It will be applied on enamel of teeth in the control group. The application is according the instruction for use within the indication. |
| Number of<br>Participants with<br>Rationale: | 23, rationale see statistical considerations |
| Duration of the investigation: | 6 months estimated duration for the main investigational plan (e.g. from start of screening of first participant to last participant processed and finishing the clinical investigation) 1 year 6 months of First-Participant-In until Last-Participant-Out |
| Investigation<br>Schedule: | Intervention, 4 weeks, 6 months, 12 months recall |
| Study Coordinator: | Mutlu Özcan Prof. Dr. h.c., Ph.D, University of Zurich Division of Dental Biomaterials Center of Dental Medicine Clinic of Reconstructive Dentistry Plattenstrasse 11, CH-8032, Zurich, Switzerland Mobile: E-mail: |
| Principal<br>Investigator: | Dr. Burcu Gözetici Istanbul Medipol University School of Dentistry Department of Restorative Dentistry Birlik Mah., Bahçeler Cd. No:5, 34230 Esenler Istanbul, TURKEY E-mail: |
| Investigation Site(s): | Single-centre |
| Statistical Considerations: | t-test allows a sample size of 23 patient with power of 80% at a significance level of 5%. |



Compliance Statement:

This clinical investigation will be conducted in compliance with the CIP (protocol), the current version of the Declaration of Helsinki, ISO EN 14155, ICH-GCP (as far as applicable) as well as all national legal and regulatory requirements.

## 2. Definitions, Terms, Abbreviations

ADE Adverse Device Effect. Adverse events (see below) that are

related to the MD under investigation or the comparator and to

the procedures involved.

For users or other persons this is restricted to events related to

the MD.

AE Adverse event (Art. 2 Abs 57 MDR):

Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related

to the MD.

Castor EDC Electronic data capturing (EDC) platform from the company

Castor

CE Conformité Européenne (Label on products complaint to

European Medical Device Legislation)

CER Clinical Evaluation Report
CIP Clinical Investigation Plan
CIR Clinical Investigation Report

Clinical studies Systematic investigation in one or more human subjects,

undertaken to assess the clinical performance, effectiveness or

safety of a medical device.

Note: For the purpose of this document, "clinical investigation" or "clinical trial"

are synonymous with "clinical study"

DD Device Deficiency (Art. 2 Abs 59 MDR):

Inadequacy of a medical device related to its identity, quality, durability, reliability, safety or performance, of an investigational device, including malfunction, user errors and inadequate

information supplied by the manufacturer.

The definition includes deficiencies related to the investigational

MD or the comparator MD.

(e)CRF (electronic) Case Report Form

ICH-GCP International Conference on Harmonisation – Good Clinical

Practice

IB Investigator's Brochure ICF Informed Consent Form

ISO International Organization for Standardization

MD Medical Device

Directive)

PI Principal Investigator

SAE Serious adverse event: (Art. 2 Abs 58 MDR)

Any adverse event (see definition above) that led to any of the

following:



- (a) death,
- (b) serious deterioration in the health of the subject that resulted in any of the following:
- (i) life-threatening illness or injury,
- (ii) permanent impairment of a body structure or a body function,
- (iii) hospitalization or prolongation of patient hospitalization\*,
- (iv) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
- (v) chronic disease,
- (c) foetal distress, foetal death or a congenital physical or mental impairment or birth defect.

\*Note: planned hospitalization for pre-existing condition, or a procedure required by the CIP, without a serious deterioration of the health status of the subject, is not considered an SAE Suspected Serious Device Effect.

SAE related to the MD and/or the comparator

Participants (i.e. Patients) that are included in a clinical investigation.

SADE Subjects



# 3. Study Schedule

| Study Periods | Screening,<br>Patient<br>information | Treatment,<br>Intervention<br>(Enrolment) | Follow-Up (Recall) | | |
|---|---|---|---|---|---|
| Visit | 1 | 2 x | 3 | 4 | 5 |
| Time (hour [h],<br>day [d], week<br>[wk], month [mt]) | 12 mt | 1 h | 4 w | 6 mt | 12 mt |
| Patient<br>Information | X | | | | |
| Informed<br>Consent | X | | | | |
| Medical History | х | | | | |
| In- /Exclusion<br>Criteria | х | х | | | |
| Tooth<br>Examination | х | | | | |
| Vitality test | х | | | | |
| VAS for tooth sensitivity | Х | | | | |
| Intraoral pictures | | Х | Х | X | Х |
| Recording<br>ICDAS and<br>Nyvad scores | | x | X | X | X |
| Professional cleaning of tooth suface | | Х | | | |
| QrayCam Pro<br>measurement | | x | x | x | x |
| Adverse events (incl. SAE) | Х | Х | х | х | x |
| Concomitant medications | Х | Х | Х | Х | Х |